CLINICAL TRIAL: NCT00521612
Title: Prospective Randomised Controled Trial: Comparison of Volatile Anaesthetics Sevoflurane vs. Isoflurane for Low-Flow General Anaesthesia for Abdominal Surgery
Brief Title: Sevoflurane vs. Isoflurane for Low-Flow General Anaesthesia for Abdominal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital Dubrovnik (Other)
Responsible Party: Ante Crncevic, MD, MSc., General Hospital Dubrovnik
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 75736
Record Dates: First submitted 2007-08-27; First posted 2007-08-28 (Estimated); Last update posted 2008-01-07 (Estimated); Status verified 2007-12

CONDITIONS: Anaesthesia
Keywords: sevoflurane; isoflurane; anaesthesia
MeSH Terms: interventions — Sevoflurane; Isoflurane

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Sevoflurane group, experimental group
  Interventions: Drug: sevoflurane
- B (Active Comparator): Isoflurane group, control group
  Interventions: Drug: isoflurane

INTERVENTIONS:
Drug: sevoflurane — Volatile anaesthetic sevoflurane 1 MAC (2,0 vol%) will be administer to the patients in the form of gas (via respiration). First 20 minutes of anaesthesia will be period of saturation of the body with anaesthetic sevoflurane. After 20 minutes the depth of anaesthesia will be titrated with level of anaesthetic sevoflurane. Change will be +10 % of sevoflurane MAC (0,2 vol%) for every change of signs that indicate shallow anaesthesia. Change will be -10 % of sevoflurane MAC (0,2 vol%) for every change of signs that indicate too deep anaesthesia. Measuring points will be every 5 minutes during surgery.
  Other Names: Sevorane
  Arms: A
Drug: isoflurane — Volatile anaesthetic isoflurane 1 MAC (1,2 vol%) will be administer to the patients in the form of gas (via respiration). First 20 minutes of anaesthesia will be period of saturation of the body with anaesthetic isoflurane. After 20 minutes the depth of anaesthesia will be titrated with level of anaesthetic isoflurane. Change will be +10 % of isoflurane MAC (0,12 vol%) for every change of signs that indicate shallow anaesthesia. Change will be -10 % of isoflurane MAC (0,12 vol%) for every change of signs that indicate too deep anaesthesia. Measuring points will be every 5 minutes during surgery.
  Other Names: Forane
  Arms: B

SUMMARY:
Two groups of patients are going to have abdominal surgery with low-flow general anaesthesia. Group A (sevoflurane group, experimental group) will use volatile anaesthetic sevoflurane. Group B (isoflurane group, control group) will use volatile anaesthetic isoflurane. It will be observed differences between volatile anaesthetic sevoflurane and volatile anaesthetic isoflurane for providing low-flow general anaesthesia for abdominal surgery. Duration of this randomised controled trial will be approximately 2 months. Estimated sample size will be 82 persons (41 in sevoflurane group and 41 in isoflurane group).

DETAILED DESCRIPTION:
Two groups of patients are going to have abdominal surgery with low-flow general anaesthesia.

Group A (sevoflurane group, experimental group) Patients will receive midazolam for premedication 45 minutes before surgery. Dose is 0,08 mg/kg i.m. Patients will be preoxygenated with 100 % oxygen with oxygen flow of 7,5 L/min. When peripheral blood saturation reach 100 %, the induction of general anaesthesia will start. For induction patients will get anaesthetic thiopental 4,5 mg/kg i.v., analgetic fentanyl 3 mcg/kg i.v. and muscle relaxant vecuronium 0,1 mg/kg i.v. After 90 seconds patients will be intubated. After intubation anaesthetic gases will be switched on. Oxygen and nitrous oxide (50:50 %) and volatile anaesthetic sevoflurane 1 MAC (2,0 vol%). Patients will be ventilated by anaesthetic device. Intermittent positive pressure ventilation (IPPV) tidal volume 8 mL/kg, respiratory rate 12 times per minute, flow will be 1 L/min. First 20 minutes of anaesthesia will be period of saturation of the body with anaesthetic sevoflurane. After 20 minutes the depth of anaesthesia will be titrated with level of anaesthetic sevoflurane. Change will be +10 % of sevoflurane MAC (0,2 vol%) for every change of signs that indicate shallow anaesthesia. Change will be -10 % of sevoflurane MAC (0,2 vol%) for every change of signs that indicate too deep anaesthesia. Signs that show the depth of anaesthesia are: arterial blood pressure (systolic, diastolic and mean), heart rate and bispectral index (BIS). Measuring points will be every 5 minutes during surgery. The goal is to provide the values of this vital signs within normal physiology ranges. Analgetic fentanyl will be repeated every 45 minutes in the dose of 0,8 mcg/kg i.v. Muscle relaxant vecuronium will be repeated in the dose of 0,5 mg/kg i.v. when train of four (TOF) shows score 30 % or higher. It will also be measured (every 5 minutes): inspiratory and expiratory concentration of sevoflurane, saturation of the blood with oxygen and level of end-tidal carbon dioxide. At the end of surgery, begins awakening from general anaesthesia. All anaesthetic gases will be switched off. Patients will be ventilated manually with 100 % oxygen with oxygen flow of 7,5 L/min. Every patient will get atropin 1 mg + neostigmine 2,5 mg i.v. for decurarization. Measuring points will be: start of awakening, extubation and discharge from operating theatre. It will be measured: arterial blood pressure (systolic, diastolic and mean), heart rate, inspiratory and expiratory concentration of sevoflurane, saturation of the blood with oxygen, level of end-tidal carbon dioxide, BIS and TOF. During surgery each patient will get i.v. infusion 2000 mL of sodium chloride 0.9 %.

Group B (isoflurane group, control group) Patients will receive midazolam for premedication 45 minutes before surgery. Dose is 0,08 mg/kg i.m. Patients will be preoxygenated with 100 % oxygen with oxygen flow of 7,5 L/min. When peripheral blood saturation reach 100 %, the induction of general anaesthesia will start. For induction patients will get anaesthetic thiopental 4,5 mg/kg i.v., analgetic fentanyl 3 mcg/kg i.v. and muscle relaxant vecuronium 0,1 mg/kg i.v. After 90 seconds patients will be intubated. After intubation anaesthetic gases will be switched on. Oxygen and nitrous oxide (50:50 %) and volatile anaesthetic isoflurane 1 MAC (1,2 vol%). Patients will be ventilated by anaesthetic device. Intermittent positive pressure ventilation (IPPV) tidal volume 8 mL/kg, respiratory rate 12 times per minute, flow will be 1 L/min. First 20 minutes of anaesthesia will be period of saturation of the body with anaesthetic isoflurane. After 20 minutes the depth of anaesthesia will be titrated with level of anaesthetic isoflurane. Change will be +10 % of isoflurane MAC (0,12 vol%) for every change of signs that indicate shallow anaesthesia. Change will be -10 % of isoflurane MAC (0,12 vol%) for every change of signs that indicate too deep anaesthesia. Signs that show the depth of anaesthesia are: arterial blood pressure (systolic, diastolic and mean), heart rate and bispectral index (BIS). Measuring points will be every 5 minutes during surgery. The goal is to provide the values of this vital signs within normal physiology ranges. Analgetic fentanyl will be repeated every 45 minutes in the dose of 0,8 mcg/kg i.v. Muscle relaxant vecuronium will be repeated in the dose of 0,5 mg/kg i.v. when train of four (TOF) shows score 30 % or higher. It will also be measured (every 5 minutes): inspiratory and expiratory concentration of isoflurane, saturation of the blood with oxygen and level of end-tidal carbon dioxide. At the end of surgery, begins awakening from general anaesthesia. All anaesthetic gases will be switched off. Patients will be ventilated manually with 100 % oxygen with oxygen flow of 7,5 L/min. Every patient will get atropin 1 mg + neostigmine 2,5 mg i.v. for decurarization. Measuring points will be: start of awakening, extubation and discharge from operating theatre. It will be measured: arterial blood pressure (systolic, diastolic and mean), heart rate, inspiratory and expiratory concentration of isoflurane, saturation of the blood with oxygen, level of end-tidal carbon dioxide, BIS and TOF. During surgery each patient will get i.v. infusion 2000 mL of sodium chloride 0.9 %.

Duration of this randomised controled trial will be approximately 2 months. Estimated sample size will be 82 persons (41 in sevoflurane group and 41 in isoflurane group).

ELIGIBILITY:
Inclusion Criteria:

* Every patient who is older than 18 years and who volunteer for this randomised controled trial and give written permission for participating in this study.
* Patients ASA I or ASA II.
* Only patients who need elective abdominal surgery (not urgent surgery).
* Patient body mass between 60 and 100 kg.

Exclusion Criteria:

* Patients younger than 18 years
* Patients ASA III and higher
* Patients who need urgent abdominal surgery
* Patients allergic to anaesthetics
* Pregnant women
* Patients with neuromuscular diseases; and
* Persons with epidural analgesia catheter.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2007-09; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Differences between volatile anaesthetic sevoflurane and volatile anaesthetic isoflurane for providing low-flow general anaesthesia for abdominal surgery. | approximately time for this trial is about 2 months

SECONDARY OUTCOMES:
Differences in awakening patients from low-flow general anaesthesia provided by sevoflurane and isoflurane. | approximately time for this trial is about 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Ante Crncevic, MD, MSc., Principal Investigator — specialist in anaesthesiology and intensive care medicine; Zoran Dogas, MD, PhD., Study Chair — Professor of Neuroscience, University of Split, School of Medicine
Locations (1):
- General Hospital Dubrovnik, Dubrovnik, Croatia

REFERENCES:
- [Background] Mahajan VA, Ni Chonghaile M, Bokhari SA, Harte BH, Flynn NM, Laffey JG. Recovery of older patients undergoing ambulatory anaesthesia with isoflurane or sevoflurane. Eur J Anaesthesiol. 2007 Jun;24(6):505-10. doi: 10.1017/S0265021506001980. Epub 2007 Jan 4. PMID 17202009
- [Background] Venkatesh BG, Mehta Y, Kumar A, Trehan N. Comparison of sevoflurane and isoflurane in OPCAB surgery. Ann Card Anaesth. 2007 Jan;10(1):46-50. doi: 10.4103/0971-9784.37924. PMID 17455408
- [Background] Seitsonen ER, Yli-Hankala AM, Korttila KT. Similar recovery from bispectral index-titrated isoflurane and sevoflurane anesthesia after outpatient gynecological surgery. J Clin Anesth. 2006 Jun;18(4):272-9. doi: 10.1016/j.jclinane.2005.12.005. PMID 16797429
- [Background] Sakai EM, Connolly LA, Klauck JA. Inhalation anesthesiology and volatile liquid anesthetics: focus on isoflurane, desflurane, and sevoflurane. Pharmacotherapy. 2005 Dec;25(12):1773-88. doi: 10.1592/phco.2005.25.12.1773. PMID 16305297
- [Background] Nakayama M, Kanaya N, Edanaga M, Namiki A. Hemodynamic and bispectral index responses to tracheal intubation during isoflurane or sevoflurane anesthesia. J Anesth. 2003;17(4):223-6. doi: 10.1007/s00540-003-0186-4. PMID 14625708
- See also: Web site of General Hospital Dubrovnik — http://www.bolnica-du.hr